CLINICAL TRIAL: NCT05869630
Title: Investigation Into the Effects of Exercise on microRNA Expressions in Patients With Knee Osteoarthritis
Brief Title: Exercise on microRNA in Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OA_exercise_microrna
Record Dates: First submitted 2023-05-06; First posted 2023-05-22 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Osteoarthritis, Knee; Epigenetic Disorder; Quality of Life; Depression; Pain
Keywords: Osteoarthritis; Epigenetic Disorder; Quality of Life; Depression; Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Depression; Pain; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Prospective Cohort Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Group (Experimental): A total of 30 knee OA patients and 30 age/sex-matched healthy volunteers were included in the exercise and control groups. Exercises were performed twice a week under supervision and once a week as home program for eight weeks. Before and after exercise treatment, peripheral venous blood samples were taken from both groups. miRNA-146a, miRNA-155, miRNA-221-3p and miRNA-145 gene expressions were studied with the Real-time PCR method. miRNA-146a, miRNA-155, and miRNA-221-3p, miRNA-145 gene expressions were studied with the Real-time PCR method. The pain was evaluated with the Numeric Rating Scale (NRS), functional status with Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), depression level with the Beck Depression Inventory (BDI), and quality of life with Short Form-36 (SF-36).
  Interventions: Other: Exercise Programme; Other: Experiments

INTERVENTIONS:
Other: Exercise Programme — All patients were informed about knee OA, joint protection principles, and the exercise effects on knee OA before treatment. The exercises were supervised by a physiotherapist for 30 minutes twice a week and once a week as a home program. The exercise program consisted of a warm-up, strengthening knee extensors and lower extremity stretching exercises. Firstly, quadriceps isometric and adductor isometric (roll tightening) exercises, hamstring stretching, quadriceps stretching, and gastrocnemius stretching were applied. Then, hip flexion-extension-abduction-adduction, and knee extension while sitting were applied with exercise bands. Strengthening exercises were composed of three sets with 10 repetitions. Stretching exercises were performed 10 repetitions for 10 seconds.
Other: Experiments — The total RNA was isolated from peripheral blood samples taken from patients and the control group by applying the protocol of the manufacturer (LucigenMasterPure™ Complete DNA and RNA Purification Kit, USA). The total RNA was isolated in three steps: Lysis stage of the whole blood samples, precipitation of nucleic acids and precipitation of total RNA. The purity and concentration of the isolated total RNA samples were measured with the spectrophotometer (Thermo Fischer) device. The samples were stored at -80°C until the next step. To determine the microRNA expression levels; firstly, conjugate DNA (cDNA) was synthesized from total RNA samples according to the manufacturer's protocol. Whether the desired region reproduced in the reaction and whether there were primer dimers were checked by adding a melting curve step. In addition, blood samples of 30 age-sex matched healthy volunteers were compared.

SUMMARY:
The present study is a prospective cohort study. This study will be conducted to determine the change in miRNA levels with exercise in knee Osteoarthritis (OA) patients. The main questions that the study aims to answer are:

Question 1: Does exercise therapy affect microrna expressions in patients with knee osteoarthritis?

Question 2: Does exercise therapy affect quality of life, pain, functional status and depression level in patients with knee osteoarthritis?

Participants; demographic information such as age, height, weight will be questioned. Exercises will performed twice a week under supervision and once a week as home program for eight weeks. Before and after exercise treatment, peripheral venous blood samples will taken from both groups. miRNA-146a, miRNA-155, miRNA-221-3p and miRNA-145 gene expressions will studied with the real-time PCR (polymerase chain reaction) method. miRNA-146a, miRNA-155, and miRNA-221-3p, miRNA-145 gene expressions will studied with the Real-time PCR method. The pain will evaluated with the Numeric Rating Scale (NRS), functional status with Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), depression level with the Beck Depression Inventory (BDI), and quality of life with Short Form-36 (SF-36).

DETAILED DESCRIPTION:
Osteoarthritis is a degenerative disease causing joint pain, stiffness, and limitation of motion with loss of cartilage, osteophyte development, subchondral sclerosis, changes in the joint capsule and synovial membrane as a result of the disruption of genetic, biomechanical, and biochemical balances. Pharmacological treatments of osteoarthritis include simple analgesics, non-steroidal anti-inflammatory drugs, opioids and topical analgesics. Patient education, self-management programs, exercise, weight loss, assistive devices and lifestyle changes are non-pharmacological treatment methods.Exercise is one of the basic elements of the treatment modality. The purpose of the exercise; to relieve symptoms and improve muscle strength around joints. It is aimed to increase the quality of life with the adaptation of individuals to exercise.

miRNA, one of the small non-coding RNA subunits, is responsible for the modulation of protein-coding genes as a result of post-transcriptional repression. miRNA play an active role in many biological events such as cellular differentiation, apoptosis, proliferation, erythropoiesis, fibrosis and angiogenesis. Due to the role of miRNAs in normal development and diseases, it is thought that they will be a new biomarker for therapeutic purposes in the future. It was found that miRNAs play a key role in physiological conditions e.g. skeletal muscle hypertrophy, mitochondrial biogenesis, vascular angiogenesis, and metabolic events when combined with exercise. The identification of miRNAs that change in circulation with exercise is important in terms of providing new data on the physiological adaptation of exercise. In recent years, a large number of miRNAs have been identified in osteoarthritic tissues, which is important in terms of the regulation of gene expressions related to the pathogenesis of OA. OA-specific miRNA expressions is necessary for early diagnosis and treatment of OA as well as for monitoring the progression of the disease. It has been reported that miRNA-146a is intensely expressed in OA tissue and its expression is induced by inflammatory cytokines. MiRNA-145 is associated with chondrocyte homeostasis and is thought to be involved in the degradation of the extracellular matrix. MiRNA-155 is a miRNA that has a role in the development and regulation of innate and acquired immunity, and its expression is increased in tissues with OA compared to healthy tissue. It has an important role in hematopoiesis. MiRNA-221-3p was found to be associated with chondrocyte proliferation, gene expression, matrix degradation and apoptosis.

In this study it was aimed to determine the changes in miRNA levels of knee OA patients with exercise.

ELIGIBILITY:
Inclusion Criteria:

* Having Kellgren-Lawrence grade 2 or grade 3 knee OA
* Body mass index (BMI) between 20-35.

Exclusion Criteria:

* Rheumatoid Arthritis,
* Having knee replacement surgery,
* Intra-articular injection in the last six months,
* Usage of opioid analgesics or corticosteroids,
* Being under severe pain (VAS>7),
* Pregnancy,
* Having cardiovascular disease,
* Stroke and chronic obstructive pulmonary disease (COPD).

Ages: 38 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2020-06-17 (Actual)

PRIMARY OUTCOMES:
Pre-Treatment Gene Expressions of microRNA for Treatment Group | Baseline
  By examining the expression level of RNA, U6 small nuclear 1 (human) as a control gene, it is decided whether the expression levels of microRNAs are expressed up or down.
Post-Treatment Gene Expressions of microRNA for Treatment Group | Through study completion, an average of 2 months.
  By examining the expression level of RNA, U6 small nuclear 1 (human) as a control gene, it is decided whether the expression levels of microRNAs are expressed up or down.
Gene Expressions of microRNA for Healthy Control Group | Baseline
  By examining the expression level of RNA, U6 small nuclear 1 (human) as a control gene, it is decided whether the expression levels of microRNAs are expressed up or down.
Pre-Treatment Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) for Treatment Group | Baseline
  WOMAC was used to evaluate functional status. There are a total of 24 questions on pain, morning stiffness and physical function.
  0 points means 'not at all', 1 point means 'mild', 2 points 'moderate', 3 points 'severe', 4 points 'very severe'.
  The total score is between 0 and 100, and a low score means that the individual is in good health.
Post-Treatment Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) for Treatment Group | At the beginning of the intervention and through study completion, an average of 2 month
  WOMAC was used to evaluate functional status. There are a total of 24 questions on pain, morning stiffness and physical function.
  0 points means 'not at all', 1 point means 'mild', 2 points 'moderate', 3 points 'severe', 4 points 'very severe'.
  The total score is between 0 and 100, and a low score means that the individual is in good health.

SECONDARY OUTCOMES:
Short Form-36 (SF-36) | At the beginning of the intervention and through study completion, an average of 2 month
  SF-36 was used to evaluate quality of life. This questionnaire consists of eight subsections. Scoring is made between 0-100 for each of the subsections. Higher scores indicate better function and well-being.
Beck Depression Inventory (BDI) | At the beginning of the intervention and through study completion, an average of 2 month
  BDI was used to evaluate depression level. The test consists of 20 questions and each question includes 0, 1, 2, 3 points.
  takes. At the end of the test; The scores marked by the patient for each question are summed up and the depression status is evaluated according to the score. The higher the score, the higher the level of depression.
Numeric Rating Scale (NRS) | At the beginning of the intervention and through study completion, an average of 2 month
  NRS was used to pain level. A score of 0 means 'no pain' and a score of 10 means 'unbearable pain'.

CONTACTS AND LOCATIONS:
Overall Officials: Fulya Senem KARAAHMETOĞLU, M.Sc, Principal Investigator — Saglik Bilimleri Universitesi; Zeynep Betül ÖZCAN, M.Sc, Study Chair — Saglik Bilimleri Universitesi; Meltem VURAL, Prof. Dr., Study Chair — Istanbul Bakırköy Dr.Sadi Konuk Training and Research Hospita; Işıl ÜSTÜN, Dr., Study Chair — Istanbul Bakırköy Dr.Sadi Konuk Training and Research Hospita; Alev KURAL, Prof. Dr., Study Chair — Istanbul Bakırköy Dr.Sadi Konuk Training and Research Hospita; Sibel KURAŞ, M. Sc., Study Chair — Saglik Bilimleri Universitesi; Bekir ERDOĞAN, M.Sc, Study Chair — Saglik Bilimleri Universitesi; Halime Hanım PENÇE, Assoc. Prof., Study Director — Saglik Bilimleri Universitesi
Locations (1):
- Bakırköy Dr. Sadi Konuk Training and Hospital Research Hospital, Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)